CLINICAL TRIAL: NCT02714686
Title: Evaluation of a Mass Media Family Planning Campaign on the Uptake of Contraceptive Methods in Burkina Faso
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Innovations for Poverty Action (Other); Development Media International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPA-10535AA
Record Dates: First submitted 2016-02-09; First posted 2016-03-21 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Contraception; Family Characteristics; Family Size, Desired
Keywords: Fertility; Total Contraception Prevalence Rate; Family planning methods; Birth Control; Mass Media Campaign; Demand for contraception; Modern Contraception Prevalence Rate; Birth intervals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radio Mass Media Family Planning Campaign (Experimental): Clusters receive a three-year mass media campaign on family planning in an attempt to reduce cognitive barriers to contraception
  Interventions: Behavioral: Radio Mass Media Family Planning Campaign
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Radio Mass Media Family Planning Campaign — Short daily spots, weekly interactive shows, testimonies, and interviews with experts and community leaders on contraception and family planning
  Arms: Radio Mass Media Family Planning Campaign

SUMMARY:
In this experiment, the investigators will study the effect of a mass media family planning campaign on contraception related behavior. The study takes place in Burkina Faso, a country with an average of six children born to each woman, and a modern contraceptive prevalence rate (mCPR) estimated at 15% in 2010 at the national level, as per the Demographic Health Survey (DHS) 2010 report on Burkina Faso.

The aim of this study is to provide robust evidence on the efficiency and cost-effectiveness of an intense three-year mass media campaign focused on family planning. The campaign will diffuse messages about the financial and health benefits of family planning, and information on the different types, sources, advantages, and disadvantages of different contraceptive methods. The study will target women at the age of reproduction in rural areas of Burkina Faso to measure the effect of the intervention on total and modern contraceptive prevalence rates, perceptions of family planning, contraception-related behavior, and general gender norms.

Burkina Faso is an ideal place to evaluate the impact of a radio campaign because a high percentage of the rural population listens to local radio which is in the local language. Radio station areas are distinct because they target very local languages and their reach is limited by government decree, which allows for the implementation of a randomized control trial.

DETAILED DESCRIPTION:
Development Media International (DMI), a non-governmental organization (NGO) that runs media campaigns to induce behavioral change in developing countries, will implement the mass media campaign in conjunction with community radio stations in rural areas of Burkina Faso. The study takes place in the coverage areas of 16 radio stations, all selected in a way to prevent overlap between coverage areas, and to have different local languages through which the campaign will be diffused. This strategy limits possible "leakages" between the treatment and the control groups. Out of the 16 clusters of radio stations, 8 will be randomly assigned to receive the media campaign, and the other 8 will be left as control.

Within each radio station cluster, only small and rural villages with no access to electricity will be sampled in order to limit access to television. The radio stations being in urban to semi-urban areas, villages that are more than 5 km away from a radio station will be excluded. Villages within radio station clusters will be randomly selected to participate in the study. A household listing survey will be conducted in all selected villages to get an exhaustive list of households and the basic information on women within each household. In addition, a village survey will be conducted with village chiefs to get a better sense of the demographics and the key figures in each village.

Based on the information provided by the listing on women at the age of reproduction, eligible women will be randomly selected to participate in the study. These women will be invited to take the baseline survey, and 3 years later, the endline survey, therefore forming a panel structure.

In addition to the listing, village, and women surveys, a clinics survey will take place to monitor the demand and supply of contraceptive methods in different areas. The clinics questionnaire will ask about contraception related behavior, including perception of family planning, usage of contraception, number of pregnancies and abortions, among other things. The investigators are also seeking administrative data from clinics within radio stations areas to examine whether distribution of contraceptive products is higher in treatment areas.

The effect of the media campaign will be analyzed based on information provided by women on how they and their partners perceive and use traditional and modern contraceptive methods, and cross-verified with information provided on demand for contraception and family planning by the clinics survey.

Qualitative research will take place prior to the launch of the campaign in order to better formulate messages that could reach the target audience.

-Data collection, reporting, and analysis:

The data collection will be conducted by Innovations for Poverty Action (IPA), and NGO specialized in conducting randomized control trials (RCTs) with presence and experience in Burkina Faso.

Data will be collected through questionnaires using Personal Digital Assistance (PDA). For the qualitative research questionnaires, answers might be recorded using paper. The surveyors might audio-record some parts of some interviews with women and health facilities using the PDAs to monitor surveying quality and performance of enumerators. The resulting datasets will be coded and clearly labeled in accordance with the information provided on the questionnaires.

Data will be collected by enumerators trained by IPA on the importance of confidentiality of the data, transparency, and accuracy of reported information. Backchecks will also be conducted to make sure that the data provided is consistent and correct. Protocols have been developed to address adverse events during data collection where enumerators go back to their supervisors and to the IPA office to address any complications. In addition, high frequency checks will be conducted whenever new data comes in to monitor the quality of data collection, and how values of different variables and missing values vary by enumerators and locations. Logic checks will be conducted to make sure that the value of variables fall within logical ranges. This allows for quick detection and correction of major outliers and high rates of attrition. Finally, all adverse events will be reported to the Massachusetts Institute of Technology's internal review board (the Committee on the Use of Humans as Experimental Subjects) as quickly as possible in accordance with the human subjects requirements.

-Sample size and minimum detectable effect:

The total sample size is approximately 8,000 women across more than 250 villages in 16 radio clusters.

To calculate this sample size, power calculations were conducted using simulations in Stata. Having two levels of clustering (region and village levels), two intracluster correlation (ICC) levels were used for power calculations, both based on the 2010 DHS data for women in Burkina Faso. The DHS data revealed a modern contraceptive prevalence rate (mCPR) of 9% among women of reproductive age (both in union and single) in rural areas and regions where the study takes place.

For these calculations, a baseline level of mCPR of 12% was assumed, therefore allowing for some increase in usage over time. Based on these numbers and calculations, the study is powered to detect a minimum of 6 percentage points increase in the mCPR.

If the assumed baseline level of mCPR is close to the actual one, power is expected to increase further as the investigators will (1) use a matched stratification on baseline levels of contraception prevalence rate at the radio station level (the level of treatment assignment), in addition to stratifying village selection on distance to health clinics, and individual selection of women on several characteristics such as education and access to a radio (2) control for baseline levels of explanatory variables and the baseline level of the outcome, and (3) use a panel structure.

It is possible, however, that the total and modern contraceptive prevalence rates are higher in the actual sample than the value assumed based on the 2010 DHS data, which could reduce power.

ELIGIBILITY:
Inclusion Criteria:

Inclusion in our study of radio station clusters on which treatment will be randomized is based on the following criteria:

* The cluster has at least one local radio station with adequate Frequency Modulation (FM) rays to cover the zone
* Different radio stations' coverage areas do not overlap with each other

The criteria for village selection is the following:

* Villages must have less than 1,500 inhabitants as per the 2006 Burkina Faso census, except in a couple of radio station clusters where villages sampled had up to 4,200 inhabitants due to the low number of small villages in them.
* The radio stations through which the campaign will be diffused, being in semi-urban or urban locations, we only include villages that are more than 5 km away from these stations
* We only consider villages with limited access to electricity
* We only consider villages less than 10 km away from a clinic as per available estimates (Geographic Institute of Burkina Faso and village chiefs)

Individual level criteria:

* We only survey women at the age of reproduction, i.e. between 15 and 49 years of age as measured by the listing

Exclusion criteria:

* No particular exclusion criteria when the inclusion criteria listed above are met.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7515 (Actual)
Dates: Start 2016-04; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in Total Contraception Prevalence Rate | Baseline and 3 years
  The percentage of women using, or whose partner is using, an effective contraceptive method out of all women at the age of reproduction in the sample ("effective" method includes all modern methods, but also some effective traditional methods, such as withdrawal)
  The investigators will look at heterogeneous treatment effects by availability of supply and by access and listenership to the radio.
Change in Modern Contraception Prevalence Rate | Baseline and 3 years
  The percentage of women using, or whose partner is using, a modern contraceptive method out of all women at the age of reproduction in the sample.
  The investigators will look at heterogeneous treatment effects by availability of supply and by access and listenership to the radio.
  All secondary outcomes listed below will eventually be analyzed only if the variables had sufficient variance.

SECONDARY OUTCOMES:
Percentage of women intending to use contraception in the future | Baseline and 3 years
Percentage of women seeking family planning advice | Baseline and 3 years
Percentage of women discussing family planning with their partners and others | Baseline and 3 years
Percentage of women who are fecund and sexually active but do not want to become pregnant but are not currently using contraception | Baseline and 3 years
Average time lapse between pregnancies | Baseline and 3 years
  Limited power to test this outcome and find significant effects
Number of unwanted pregnancies | Baseline and 3 years
  Limited power to test this outcome and find significant effects
Number of births per 1,000 women of reproductive age (if accurate population level data on total births in communities become available) | Baseline and 3 years
  Limited power to test this outcome and find significant effects
Number of family planning products delivered throughout the study period (from administrative data, if available) | Baseline and 3 years
Mean effects on survey questions relating to knowledge of contraceptive methods | Baseline and 3 years
  Variables include: knowledge of the existence, price, source, advantages, and disadvantages of different methods, including rejection of misconceptions such as contraception causing sterility or sickness
Mean effects on survey questions relating to attitudes towards contraception | Baseline and 3 years
  * Percentage of women who think that it is embarrassing to buy a contraceptive method
  * Percentage of women who think that using contraceptive methods is a sign of not trusting their partner
Mean effects on survey questions relating to knowledge of family planning | Baseline and 3 years
  * Percentage of women who know benefits of spacing births
  * Percentage of women who know benefits of delaying the age of marriage for young girls
Mean effects on survey questions relating to attitudes towards family planning | Baseline and 3 years
  * Percentage of women who think it is acceptable to talk about family planning in public (radio, schools, posters, etc.)
  * Percentage of women who think that a woman should be able to control the number of children she has during her lifetime
Mean effects on survey questions relating to women's perceptions of fertility and birth spacing | Baseline and 3 years
  * Women's perception on the ideal age at first birth (in standard deviation units from the control group)
  * Women's perception on the ideal time lapse between first and second birth (in standard deviation units from the control group)
  * Women's perception on the ideal number of children in total (in standard deviation units from the control group)
Mean effects on survey questions relating to partners' perceptions of fertility and birth spacing (as reported by women) | Baseline and 3 years
  * Partners' perception on the ideal time lapse between first and second birth (in standard deviation units from the control group)
  * Partners' perception on the ideal number of children in total (in standard deviation units from the control group)
Mean effects on survey questions relating to perceptions on gender norms | Baseline and 3 years
  * Percentage of women who think that it is better to be a man than a woman
  * Percentage of women who think that boys should have better access to resources in education
  * Percentage of women who think that men must be more educated than their wives
  * Percentage of women who think that men should have better access to consumption of meat and imported products
Mean effects on survey questions relating to behavior reflecting women empowerment | Baseline and 3 years
  * Percentage of women working or participating in a productive activity
  * Percentage of women participating in decision-making when it comes to different household expenditures
Mean effects on survey questions relating to women's subjective health and wellbeing | Baseline and 3 years
  * Percentage of women satisfied with their lives
  * Percentage of women considering themselves healthy compared to other women their age in the village
  * Percentage of women considering themselves happy compared to other women their age in the village
Mean effects on survey questions relating to domestic violence and sexual harassment | Baseline and 3 years
  * Percentage of women whose husbands / husbands' families get jealous when they walk to other men
  * Percentage of women whose husbands / husbands' families don't allow them to see their female friends
  * Percentage of women whose husbands / husbands' families insist on knowing where they are in the village at any time of the day
  * Percentage of women whose husbands / husbands' families ever threatened to harm them or their families
  * Percentage of women whose husbands / husbands' families ever destroyed their personal objects
  * Percentage of women whose husbands / husbands' families ever physically hurt them

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Glennerster, PhD, Principal Investigator — Abdul Latif Jameel Poverty Action Lab; Joanna Murray, PhD, Principal Investigator — Development Media International; Victor Pouliquen, M.A., Principal Investigator — Abdul Latif Jameel Poverty Action Lab
Locations (1):
- Innovations for Poverty Action, Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
After completion of the evaluation and publication of the study, anticipated in 2021, a de-identified version of the database will be made available to a broader audience for further academic or policy oriented studies. The datasets will contain all information collected from the surveys at baseline and endline, except for personal identifiers which will be removed to protect the identity of participants.